CLINICAL TRIAL: NCT06456385
Title: Investigate the Anti-pain Effect of Transcutaneous Auricular Vagus Nerve Stimulation (taVNS) in Patients With Chronic Post-stroke Upper Extremity Pain
Brief Title: Post-stroke Pain taVNS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00137146
Record Dates: First submitted 2024-06-04; First posted 2024-06-13 (Actual); Results first posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Stroke; Pain
MeSH Terms: conditions — Stroke; Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Auricular Neurostimulation (Active) (Active Comparator): Participants will receive auricular stimulation of both the 15Hz on cymba conchae and 100Hz on tragus.
  Interventions: Device: Transcutaneous Auricular Vagus Nerve Stimulation (taVNS)
- Auricular Neurostimulation (Sham) (Sham Comparator): Participants will receive auricular stimulation of 15Hz on their earlobe.
  Interventions: Device: Sham Auricular Stimulation

INTERVENTIONS:
Device: Transcutaneous Auricular Vagus Nerve Stimulation (taVNS) — The intervention applied is called transcutaneous auricular vagus nerve stimulation (taVNS) which administers electrical stimulation at the ear which targets the auricular branch of the vagus nerve.
  Arms: Auricular Neurostimulation (Active)
Device: Sham Auricular Stimulation — The sham auricular stimulation administers electrical stimulation at the ear lobe which has less auricular branch of the vagus nerve.
  Arms: Auricular Neurostimulation (Sham)

SUMMARY:
The purpose of this study is to explore whether a non-invasive form of ear stimulation called transcutaneous auricular vagus nerve stimulation (taVNS) can change the way participants perceive pain. Investigators will recruit up to 20 participants with chronic post-stroke upper extremity pain. The goal is to determine if there is a pain reduction after ear stimulation.

DETAILED DESCRIPTION:
In this study, investigators main goal is to establish transcutaneous auricular vagus nerve stimulation (taVNS) as an effective non-invasive neuromodulation method for analgesia of post-stroke upper extremity pain. Participants are required to have an ischemic or hemorrhagic stroke that occurred at least 6 months prior and are currently suffering upper extremity pain. Each participant will undergo an in-person visit. Participants will first finish the pain questionnaires and have quantitative sensory testing (QST) conducted to determine baseline pain thresholds. Participants will then receive 30 minutes of taVNS (either active or sham). Upon the completion of the stimulation intervention, participants will then be tested for another QST and pain questionnaires.

Aim 1: Test the safety and feasibility of taVNS in participants with chronic post-stroke upper extremity pain.

Over the last 8 years, investigators have demonstrated that taVNS is safe and feasible in several different populations in our previous studies. Specifically, investigators have demonstrated that taVNS is well tolerated and safe for participants with chronic stroke in our previous clinical trial. In this study, investigators will further verify the safety and feasibility of taVNS in the population with chronic post-stroke upper extremity pain.

Aim 2: Investigate whether taVNS can modulate pain in this population compared to sham.

In this single-visit, double-blinded, sham-controlled pilot trial, investigators will compare changes in post-stroke upper extremity pain scores and pain threshold derived from QST before and after a 30-minute taVNS intervention, as well as between active and sham taVNS. The findings will help investigators understand whether taVNS can modulate pain in this population.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80
* Have the capacity and ability to provide one's own consent in English and sign the informed consent document.
* Ischemic or hemorrhagic stroke that occurred at least 6 months prior
* Unilateral stroke lesions in the left hemisphere
* Right upper extremity pain

Exclusion Criteria:

* Primary intracerebral hematoma or subarachnoid hemorrhage
* Documented history of dementia
* Documented history of uncontrolled depression or psychiatric disorder
* Uncontrolled hypertension despite treatment, specifically SBP (Systolic Blood Pressure) / DBP (Diastolic Blood Pressure) >=180/100mmHg
* Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2024-06-04 (Actual); Primary Completion 2024-09-26 (Actual); Study Completion 2024-09-26 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of South Carolina Institute of Psychiatry, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Peng X, Cox SS, Baker-Vogel B, Omonije F, Tucker K, Huttig B, Sutton F, Cash N, Wood M, Kautz SA, Badran BW, Borckardt JJ. Transcutaneous Auricular Neurostimulation Modulates Pain Perception in Survivors of Stroke With Chronic Upper-Extremity Pain: A Randomized, Sham-Controlled Pilot Study. Neuromodulation. 2026 Jan 16:S1094-7159(25)01202-4. doi: 10.1016/j.neurom.2025.12.005. Online ahead of print. PMID 41543462

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Auricular Neurostimulation (Active) | Auricular Neurostimulation (Sham)
Started | 7 | 8
Completed | 7 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Auricular Neurostimulation (Active) | Auricular Neurostimulation (Sham) | Total
Number analyzed (Participants) | 7 | 8 | 15
Age, Continuous [Mean (Standard Deviation); unit: year] | 51.43 (9.88) | 61.38 (8.43) | 56.73 (10.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 10
  Male | 1 | 4 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 3 | 8
  White | 1 | 5 | 6
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
QST Thermal Pain Threshold [Mean (Standard Deviation); unit: Celsius] — Population: One participant from the sham group did not complete the QST procedure correctly and was therefore excluded from the analysis.
  Celsius
    number analyzed (Participants) | 7 | 7 | 14
    (all) | 40.59 (4.51) | 43.01 (2.44) | 41.8 (3.75)
Subject Pain Rating [Mean (Standard Deviation); unit: scale 0-10] — Population: One participant from the sham group did not complete the QST procedure correctly and was therefore excluded from the analysis.
  scale 0-10
    number analyzed (Participants) | 7 | 7 | 14
    (all) | 4.57 (2.23) | 4.14 (2.61) | 4.36 (2.34)

OUTCOME MEASURES:

1. Primary Outcome: Thermal Pain Threshold
Description: Using a quantitative sensory testing paradigm, the investigators will systematically determine information on thermal pain tolerance thresholds (degrees celsius) using a 30 × 30 mm thermode attached to the left forearm of participants.
Time Frame: assessed during and immediately after the single 30-minute taVNS session, Post 30-minute taVNS reported
Measure: Mean (Standard Deviation); unit: Celsius
Arm/Group | Auricular Neurostimulation (Active) | Auricular Neurostimulation (Sham)
Number analyzed (Participants) | 7 | 7
Celsius | 41.84 (5.14) | 42.51 (2.66)

2. Secondary Outcome: Subjective Pain Ratings
Description: Participants will rate their post-stroke upper extremity pain intensity before and after the taVNS using a standard numeric pain rating scale (from minimum 0 to maximum 10, higher scores mean more pain).
Time Frame: assessed during and immediately after the single 30-minute taVNS session, Post 30-minute taVNS reported
Measure: Mean (Standard Deviation); unit: Scale 0-10
Arm/Group | Auricular Neurostimulation (Active) | Auricular Neurostimulation (Sham)
Number analyzed (Participants) | 7 | 7
Scale 0-10 | 4.00 (2.45) | 3.57 (2.30)

ADVERSE EVENTS:
Time Frame: up to 3 months.
Arm/Group | Auricular Neurostimulation (Active) | Auricular Neurostimulation (Sham)
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/8
Other Adverse Events (participants affected / at risk) | 0/7 | 0/8

LIMITATIONS AND CAVEATS:
This study was an early proof-of-concept pilot trial designed to establish safety and feasibility for tAN in individuals with chronic PSP. This study has a relatively small sample size, and future studies should be adequately powered to more clearly determine the clinical efficacy of tAN.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2024-06-28): https://cdn.clinicaltrials.gov/large-docs/85/NCT06456385/Prot_001.pdf